CLINICAL TRIAL: NCT03380013
Title: Pilot Study Assessing the Effect of Osteopathic Manipulative Treatment (OMT) on Length of Stay in Infants With Neonatal Encephalopathy After Therapeutic Hypothermia
Brief Title: OMT to Improve Feeding After Hypothermia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Responsible Party: Principal Investigator, Alexa Craig, Neonatal and Pediatric Neurologist, MaineHealth
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB 1134889-1
Record Dates: First submitted 2017-11-07; First posted 2017-12-20 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Neonatal Encephalopathy; Feeding; Difficult, Newborn
Keywords: hypothermia treatment; OMT in infants
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: Infants recruited for this study are treated with OMT upon completion of hypothermia. They are compared 1:3 with matched historical controls.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMT group (Experimental): Osteopathic Manipulative Therapy (OMT); two treatments between day 4 and 7 of life
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — Each neonate will have a structural exam completed assessing each body region (head, cervical, thoracic, lumbar, sacral, pelvic, rib cage, and abdominal regions) for underlying somatic dysfunctions prior to each treatment. The specific OMT techniques used will be left to the discretion of the treating physician and will not be based on a predetermined protocol. Treatment techniques will consist of myofascial release, balanced ligamentous tension, balanced membranous tension, and osteopathy in the cranial field. Total treatment time will be 15 minutes. The features of the osteopathic structural exam which will be recorded on paper by the treating physician at the time of the evaluation. The paper will be marked only with the research identifier.

SUMMARY:
The goal of this study is to determine if infants with neonatal encephalopathy will achieve full oral feeds faster after therapeutic hypothermia has completed if they are treated with osteopathic manipulative treatment. The treated infants will be compared to matched historical controls.

DETAILED DESCRIPTION:
Infants affected by neonatal encephalopathy (NE) have been shown to have better survival rates and improved long term neurodevelopment following treatment with therapeutic hypothermia. However, a barrier to hospital discharge for these infants is a successful transition from gavage to either breast or bottle feeding.

Often, the factor delaying hospital discharge is slow transition to full oral feeds. Osteopathic manipulative treatment (OMT) helps to effectively stabilize and regulate the autonomic nervous system as well as the cranial nerves important in the sucking and latching reflexes, which may in turn help to ease the transition to full oral feeding. We hypothesize that infants who receive OMT will accelerate the transition to full oral feeds, thus decreasing their overall length of hospitalization compared to historical matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Neonate > 37 weeks gestational age at birth
* Neonate been diagnosed with neonatal encephalopathy or hypoxic ischemic encephalopathy and treated with therapeutic hypothermia
* Neonate with mild to moderate encephalopathy
* EEG without seizure activity
* Brain MRI without basal ganglia injury

Exclusion Criteria:

* Neonate < 37 weeks gestational age at birth
* Neonate with severe encephalopathy (as defined by Sarnat)
* EEG demonstrated seizure activity or evidence of status epilepticus during therapeutic hypothermia treatment
* Brain MRI demonstrating moderate or severe basal ganglia injury
* Neonate affected by neonatal abstinence syndrome (NAS)
* Neonate affected by intrauterine growth restriction (IUGR)
* Neonate born with major congenital anomalies (i.e., cleft palate)
* Prenatal history of maternal insulin dependent gestational or type 1 diabetes
* Moribund status (i.e., infants unlikely to benefit from or are not responsive to aggressive life support)

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Total hospital length of stay | 4-6 weeks
  Assess the effect of OMT on total hospital length of stay. We will compare infants treated with OMT 1:3 with matched historical controls.

SECONDARY OUTCOMES:
Number of days until full oral feeding is achieved | 4-6 weeks
  Assess the effect of OMT on the number of days until full oral feeding is achieved.
Patterns of somatic dysfunction | 4-6 weeks
  We will perform an osteopathic structural exam before and after treatment while recording the specific somatic dysfunctions observed within the medical record. We will then use these notes to perform a qualitative analysis of patterns of somatic dysfunction specific to the craniosacral mechanism before and after OMT.

CONTACTS AND LOCATIONS:
Overall Officials: Alexa Craig, MD, Principal Investigator — MaineHealth
Locations (1):
- Maine Medical Center, Portland, Maine, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobs SE, Berg M, Hunt R, Tarnow-Mordi WO, Inder TE, Davis PG. Cooling for newborns with hypoxic ischaemic encephalopathy. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD003311. doi: 10.1002/14651858.CD003311.pub3. PMID 23440789
- [Background] Henley CE, Ivins D, Mills M, Wen FK, Benjamin BA. Osteopathic manipulative treatment and its relationship to autonomic nervous system activity as demonstrated by heart rate variability: a repeated measures study. Osteopath Med Prim Care. 2008 Jun 5;2:7. doi: 10.1186/1750-4732-2-7. PMID 18534024
- [Background] Inder TE. Pediatrics: predicting outcomes after perinatal brain injury. Nat Rev Neurol. 2011 Sep 13;7(10):544-5. doi: 10.1038/nrneurol.2011.142. No abstract available. PMID 21912407
- [Background] Frymann V. Relation of disturbances of craniosacral mechanisms to symptomatology of the newborn: study of 1,250 infants. J Am Osteopath Assoc. 1966 Jun;65(10):1059-75. No abstract available. PMID 5178520
- [Background] Cerritelli F, Pizzolorusso G, Ciardelli F, La Mola E, Cozzolino V, Renzetti C, D'Incecco C, Fusilli P, Sabatino G, Barlafante G. Effect of osteopathic manipulative treatment on length of stay in a population of preterm infants: a randomized controlled trial. BMC Pediatr. 2013 Apr 26;13:65. doi: 10.1186/1471-2431-13-65. PMID 23622070

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT03380013/Prot_SAP_000.pdf